CLINICAL TRIAL: NCT06937437
Title: Effects of Tele Speech Therapy on the Treatment of Stammering in Adults Who Stutter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0664
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stammering
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele therapy (Experimental): The experimental group will be given teletherapy, total number of 2 sessions per week, each participant comprising 30 minutes.
  Interventions: Other: Teletherapy
- Traditionally speech therapy (Active Comparator): Traditional therapy will be given a total of 2 sessions per week to each participant, comprised of 30 minutes
  Interventions: Other: Traditionally speech therapy

INTERVENTIONS:
Other: Teletherapy — A teletherapy patient presenting with stammering (stuttering) is a person receiving speech therapy remotely, using technology like video conferencing, to address speech fluency difficulties, often including repetitions, prolongations, or blocks in speech.
  Arms: Tele therapy
Other: Traditionally speech therapy — This type of intervention is traditional speech therapy that will be given to stammering adults, to address speech fluency difficulties, often including repetitions, prolongations, or blocks in speech.
  Arms: Traditionally speech therapy

SUMMARY:
The aim of the study is to determine the effectiveness of telespeech therapy on the treatment of stammering.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Adults With stuttering 15 to 40 years according to WHO criteria

Exclusion Criteria:

- Stammering with any comorbid are excluded eg. Visual and Hearing Impairment

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Stuttering Severity Instrument - Fourth Edition (SSI4) | Base line and 6 weeks
  The Stuttering Severity Instrument-Fourth Edition (SSI-4) is a norm-referenced assessment used to quantify stuttering severity in children and adults, measuring frequency, duration, physical concomitants, and the naturalness of speech.
  The total score measures the overall severity of the individual's stuttering disorder. The examiner adds scores from the frequency, duration, and physical concomitants sections to obtain the severity score and percentile rank. These are calculated using the tables within the record form. These tables also convert scores to a severity equivalent, which ranges from "very mild" to "very severe".
  It has a total score range of 0 to 20 for physical concomitants, and 2 to 18 for frequency and duration. The total score for the entire instrument is the sum of these three scores, making the overall range up to 20 + 18 + 18 = 56.

CONTACTS AND LOCATIONS:
Overall Officials: Mamona Riaz, M.S, Principal Investigator — Riphah International University
Locations (1):
- Muaz Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Månsson H. Childhood stuttering: Incidence and development. Journal of fluency disorders. 2000;25(1):47-57.
- [Background] Eslami Jahromi M, Ahmadian L, Bahaadinbeigy K. The effect of tele-speech therapy on treatment of stuttering. Disabil Rehabil Assist Technol. 2022 Jan;17(1):34-39. doi: 10.1080/17483107.2020.1754475. Epub 2020 Apr 17. PMID 32299263